CLINICAL TRIAL: NCT00998517
Title: Comparison of a Novel Fortified Blended Flour to Ready-to-use Supplemental Foods for the Treatment of Moderate Acute Malnutrition in Rural Malawian Children: a Randomized, Investigator-blinded, Clinical Effectiveness Trial
Brief Title: Effectiveness Comparison of Three Supplementary Foods in the Treatment of Moderate Acute Malnutrition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SOYA2009
Record Dates: First submitted 2009-10-19; First posted 2009-10-20 (Estimated); Results first posted 2014-05-12 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-04

CONDITIONS: Malnutrition
Keywords: Malnutrition; Supplemental Food; CSB++; Supplementary Plumpy
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Who Masked: Investigator

ARMS (3):
- Soy/peanut fortified spread (Active Comparator)
  Interventions: Dietary Supplement: Soy/peanut fortified spread
- Milk fortified corn/soy blend (Experimental)
  Interventions: Dietary Supplement: Milk fortified corn/soy blend
- Supplementary Plumpy® (Active Comparator)
  Interventions: Dietary Supplement: Supplementary Plumpy®

INTERVENTIONS:
Dietary Supplement: Soy/peanut fortified spread — 75kcal/kg/day
  Arms: Soy/peanut fortified spread
Dietary Supplement: Milk fortified corn/soy blend — 75 kcal/kg/day
  Arms: Milk fortified corn/soy blend
Dietary Supplement: Supplementary Plumpy® — 75 kcal/kg/day
  Arms: Supplementary Plumpy®

SUMMARY:
The purpose of this study is to compare the recovery rates of moderately malnourished Malawian children treated with either milk-enriched corn/soy blend, soy/peanut fortified spread or a commercially produced ready-to-use therapy food.

ELIGIBILITY:
Inclusion Criteria:

* WHZ <-2 but >-3 without bilateral pedal edema
* Reside within 7 kilometers of study site.

Exclusion Criteria:

* Not permanent resident in vicinity of study site.
* Severe chronic illness such as cerebral palsy.
* History of peanut allergy or anaphylaxis resulting from any food.
* Receiving other supplementary food or participating in other research.

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2712 (Actual)
Dates: Start 2009-10; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Manary, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- University of Malawi College of Medicine, Blantyre, Malawi

REFERENCES:
- [Derived] Trehan I, Banerjee S, Murray E, Ryan KN, Thakwalakwa C, Maleta KM, Manary MJ. Extending supplementary feeding for children younger than 5 years with moderate acute malnutrition leads to lower relapse rates. J Pediatr Gastroenterol Nutr. 2015 Apr;60(4):544-9. doi: 10.1097/MPG.0000000000000639. PMID 25419681
- [Derived] Chang CY, Trehan I, Wang RJ, Thakwalakwa C, Maleta K, Deitchler M, Manary MJ. Children successfully treated for moderate acute malnutrition remain at risk for malnutrition and death in the subsequent year after recovery. J Nutr. 2013 Feb;143(2):215-20. doi: 10.3945/jn.112.168047. Epub 2012 Dec 19. PMID 23256140
- [Derived] LaGrone LN, Trehan I, Meuli GJ, Wang RJ, Thakwalakwa C, Maleta K, Manary MJ. A novel fortified blended flour, corn-soy blend "plus-plus," is not inferior to lipid-based ready-to-use supplementary foods for the treatment of moderate acute malnutrition in Malawian children. Am J Clin Nutr. 2012 Jan;95(1):212-9. doi: 10.3945/ajcn.111.022525. Epub 2011 Dec 14. PMID 22170366

RESULTS

PARTICIPANT FLOW:
Groups:
- Milk Fortified Corn/Soy Blend: Milk fortified corn/soy blend : 75 kcal/kg/day
- Soy/Peanut Fortified Spread: Soy/peanut fortified spread : 75kcal/kg/day
- Supplementary Plumpy®: Supplementary Plumpy® : 75 kcal/kg/day
Period: Overall Study
Arm/Group | Milk Fortified Corn/Soy Blend | Soy/Peanut Fortified Spread | Supplementary Plumpy®
Started | 888 | 906 | 918
Completed | 888 | 906 | 918
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Milk Fortified Corn/Soy Blend | Soy/Peanut Fortified Spread | Supplementary Plumpy® | Total
Number analyzed (Participants) | 888 | 906 | 918 | 2712
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 888 | 906 | 918 | 2712
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.63 (0.92) | 1.63 (0.9) | 1.61 (0.92) | 1.62 (0.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 539 | 562 | 583 | 1684
  Male | 349 | 344 | 335 | 1028
Region of Enrollment [Number; unit: participants]
  Malawi | 888 | 906 | 918 | 2712

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Nutritional Recovery
Description: Recovery is defined by weight for height Z (WHZ) score of -2 or greater using enrollment length.
  WHZ will be computed using standard WHO growth standards: http://www.who.int/childgrowth/standards/en/
Time Frame: 12 weeks or upon completion of recovery
Measure: Number; unit: participants
Arm/Group | Milk Fortified Corn/Soy Blend | Soy/Peanut Fortified Spread | Supplementary Plumpy®
Number analyzed (Participants) | 888 | 906 | 918
participants | 763 | 795 | 807

2. Primary Outcome: Number of Patients With Absence of Bilateral Pedal Pitting Edema
Time Frame: 12 weeks or recovery
Measure: Number; unit: participants
Arm/Group | Milk Fortified Corn/Soy Blend | Soy/Peanut Fortified Spread | Supplementary Plumpy®
Number analyzed (Participants) | 888 | 906 | 918
participants | 850 | 871 | 879

3. Secondary Outcome: Rate of Weight Gain
Description: This rate will be measured up to the 2nd followup visit (4 weeks) or up to the 1st followup visit (2 weeks) if the child recovered after only 2 weeks
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: g/kg/d
Arm/Group | Milk Fortified Corn/Soy Blend | Soy/Peanut Fortified Spread | Supplementary Plumpy®
Number analyzed (Participants) | 888 | 906 | 918
g/kg/d | 3.1 (2.4) | 3.4 (2.6) | 3.6 (2.8)

4. Secondary Outcome: Number of Patients With Adverse Outcomes
Description: This includes children with allergic or other adverse reactions that could be attributed to their assigned intervention food.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Milk Fortified Corn/Soy Blend | Soy/Peanut Fortified Spread | Supplementary Plumpy®
Number analyzed (Participants) | 888 | 906 | 918
participants | 0 | 0 | 0

5. Secondary Outcome: Number of Patients With Fever, Cough, and Diarrhea During the First Two Weeks of Treatment
Time Frame: 2 weeks
Measure: Number; unit: participants
Arm/Group | Milk Fortified Corn/Soy Blend | Soy/Peanut Fortified Spread | Supplementary Plumpy®
Number analyzed (Participants) | 888 | 906 | 918
participants
  diarrhea during first 2 weeks | 271 | 303 | 309
  vomiting during first 2 weeks | 89 | 127 | 124

6. Secondary Outcome: Remain Well-nourished Through 12 Months Following Successful Treatment for Moderate Acute Malnutrition (MAM)
Description: Children who were successfully treated for MAM in the primary portion of the study were followed prospectively with scheduled follow-up visits for 12 months to evaluate whether they remained well-nourished, defined as mid-upper arm circumference (MUAC) >= 12.5 cm or weight-for-height Z-score >= -2 throughout the duration of follow-up.
Time Frame: 12 months
Population: Children who successfully recovered from MAM following the standard treat-to-WHZ -2 protocol.
Measure: Number; unit: participants
Arm/Group | Milk Fortified Corn/Soy Blend | Soy/Peanut Fortified Spread | Supplementary Plumpy®
Number analyzed (Participants) | 653 | 647 | 667
participants
  well-nourished | 402 | 382 | 446
  relapsed into MAM | 110 | 117 | 107
  developed marasmus | 35 | 28 | 20
  developed kwashiorkor | 28 | 47 | 32
  died | 32 | 19 | 23
  lost to follow-up | 46 | 54 | 39

7. Secondary Outcome: Rates of Gain in Mid-upper Arm Circumference, and Length
Description: These rates will be measured up to the 2nd followup visit (4 weeks) or up to the 1st followup visit (2 weeks) if the child recovered after only 2 weeks
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: mm/d
Arm/Group | Milk Fortified Corn/Soy Blend | Soy/Peanut Fortified Spread | Supplementary Plumpy®
Number analyzed (Participants) | 888 | 906 | 918
mm/d
  MUAC gain (mm/d) | 0.13 (0.40) | 0.13 (0.43) | 0.21 (0.44)
  length gain (mm/d) | 0.13 (0.46) | 0.13 (0.44) | 0.15 (0.47)

ADVERSE EVENTS:
Arm/Group | Milk Fortified Corn/Soy Blend | Soy/Peanut Fortified Spread | Supplementary Plumpy®
Serious Adverse Events (participants affected / at risk) | 0/888 | 0/906 | 0/918
Other Adverse Events (participants affected / at risk) | 0/888 | 0/906 | 0/918

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes